CLINICAL TRIAL: NCT02203838
Title: An Open-Label, Long-Term Safety and Tolerability Study of RBP-7000 in the Treatment of Subjects With Schizophrenia
Brief Title: Long Term Study of RBP 7000 in the Treatment of Subjects With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-13-0005
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic; Schizophrenias; Risperidone; Long-acting Risperidone; Atrigel; Subcutaneous
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RBP-7000 - 120-mg dose (Experimental): RBP-7000 120-mg subcutaneous (SC) injections every 28 days for 13 doses as open-label therapy. Patients enter the study as 'roll-over' patients from study RB-US-09-0010, or de novo patients. Pre-study procedures vary for de novo patients depending on previous therapy.
  Interventions: Drug: RBP-7000

INTERVENTIONS:
Drug: RBP-7000 — 120-mg RBP-7000 dose delivered by subcutaneous injection every 28 days for a total of 13 injections (for roll-over participants, the first two injections took place under study RB-US-09-0010).
  A one-time down-titration to 90 mg RBP-7000 is permitted at the investigator's discretion should the participant have tolerability issues. Participants who received the 90-mg dose of RBP-7000 and exhibited a worsening in psychiatric symptoms could receive a one-time up-titration back to 120 mg RBP-7000 at the discretion of the investigator.
  RBP-7000 is a combination of the ATRIGEL Delivery System and risperidone. The ATRIGEL Delivery System allows for sustained-release of risperidone in a controlled manner.
  Other Names: Risperidone; Long-acting Risperidone

SUMMARY:
This is a Phase 3, open label study administering RBP-7000 in the treatment of patients with schizophrenia. Study will assess the long-term safety and tolerability of RBP-7000 subcutaneous (SC) injections in subjects with schizophrenia and to continue collecting clinical outcome data with RBP-7000 SC injections in subjects with schizophrenia using the Positive and Negative Syndrome Scale (PANSS) and Clinical Global Impression-Severity Illness (CGI-S) scale.

DETAILED DESCRIPTION:
Patients to be screened must be diagnosed with schizophrenia with a designated score based on the PANSS, as confirmed by a State, Assessability, Face, Ecological and Rule (SAFER) interview. "De novo" patients are patients who are already receiving 3- or 4-mg oral risperidone/day and will not have to complete the "run-in" or "conversion" phases (see below) and will be assigned to receive RBP-7000 after eligibility has been confirmed. Patients who completed the double-blind, placebo-controlled, efficacy study of RBP-7000 (RB-US-09-0010, NCT02109562), conducted in patients with acute schizophrenia (referred to as "roll-over" patients) will be screened.

All patients will be assigned the 120 mg dose of RBP-7000, which is subject to a one-time down-titration to 90-mg RBP-7000 for tolerability, at the investigator's discretion. Patients receiving the 90-mg dose of RBP-7000 who exhibit a worsening in psychiatric symptoms, confirmed by a total PANSS score >70 or a 20% increase in the PANSS score from the previous assessment at the 120-mg dose level (before the dose was decreased to 90 mg), can receive a one-time, up-titration back to 120-mg RBP-7000 at the discretion of the investigator.

"De novo" patients entering into the study are those patients who did not participate in study RB-US-09-0010 (NCT02109562) and are allocated into three groups with different pre-study procedures to prepare for the treatment period:

* "Run-in" patients are patients who are not already receiving oral risperidone (as no other antipsychotic medications are allowed during study participation) and will begin a 14-day run-in period by titrating up to a dose of 3 or 4 mg oral risperidone/day before the first injection of RBP-7000.
* "Conversion" patients are patients who are receiving oral risperidone doses other than 3 or 4mg/day and will begin a 7-day conversion period to achieve an oral risperidone dose level of 3 or 4-mg before the first injection of RBP-7000, only if clinically indicated.
* De novo patients taking an oral risperidone dose of 3 or 4 mg/day prestudy will (once screened/enrolled) receive the first injection of RBP-7000.

"Roll-over" patients entering into the study are patients who completed 56 days of double-blind treatment in Study RB-US-09-0010. These patients will be eligible to enter the current study provided that continuation of treatment is clinically warranted, as judged by the investigator, and that there have been no significant protocol deviations or clinically relevant adverse events (AEs) that would preclude inclusion in this study. Roll-over patients will not undergo the complete screening process and will not require either a run-in or conversion period with oral risperidone. On Day 1 of the open-label study (which is Day 57 of Study RB-US-09-0010), patients will receive their first injection (120 mg) of open label RBP-7000.

ELIGIBILITY:
Inclusion Criteria:

"De Novo" Patients

* Diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual, Edition 4, text revision (DSM-IV-TR) criteria
* Total PANSS score <=70 at the time of screening (Visit 1)
* Otherwise healthy on the basis of physical examinatIon
* Provided written informed consent

"Roll-over Patients

* Provided written consent to participate in this study
* Be considered eligible to enroll based on End of Study (EOS) (Day 57 of Study RB-US-09-0010) assessments and the medical judgment of the investigator

Exclusion Criteria:

"De Novo" Patients

* Patients taking daily oral risperidone at a dose plus/minus 6 mg/day
* Patients taking any risperidone or 9-hydroxyrisperidone long-acting injectable formulation within 120 days of study screening (Visit 1)
* Patients who have received a long-acting injectable antipsychotic within 120 days of screening (Visit 1)
* Patients with evidence or history (in the past six months prior to screening) of a significant hepatic disorder that may either compromise patient safety or interfere with the safety and/or outcome evaluation of the study drug, including:

  * Acute or chronic hepatitis, including but not limited to hepatitis B or C
  * Total bilirubin greater than 1.5 times the upper limit of normal (ULN), or
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2 times ULN
* Patients with a history of drug-induced leukopenia
* Patients with other medical conditions including, but not limited to, history of heart attack (myocardial infarction) or brain injury (traumatic injury with loss of consciousness and/or cerebrovascular accident), and clinically significant low blood pressure or arrhythmias as interpreted by the primary investigator (PI) or medically qualified sub-investigator
* Patients with epilepsy or other seizure disorders, Parkinson's disease or dementia

"Roll-over" Patients

* Patients requiring an inpatient treatment setting at the end of Study RB-US-09-0010
* Patients with an unstable medical condition developed during Study RB-US-09-0010
* Women of childbearing potential who have a positive pregnancy test at screening (Visit 1), who are pregnant or breastfeeding, seeking pregnancy, or failing to use adequate contraceptive methods during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indivior Inc., Study Director — Indivior Inc.
Locations (48):
- United States (48):
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Springdale, Arkansas
  - Comprehensive Clinical Development, Cerritos, California
  - Synergy EPIC, Escondido, California
  - Behavioral Research Specialists, Glendale, California
  - Collaborative Neuroscience Network, LLC, Long Beach, California
  - Apostle Clinical Trials, Long Beach, California
  - Pacific Research Partners, Oakland, California
  - Excell Research, Oceanside, California
  - CNRI-Los Angeles, Pico Rivera, California
  - CNRI-San Diego, San Diego, California
  - Research Center for Clinical Studies, Norwalk, Connecticut
  - Comprehensive Clinical Development-Washington DC, Washington D.C., District of Columbia
  - Florida Clinical Research Center, Bradenton, Florida
  - Innovative Clinical Research, Fort Lauderdale, Florida
  - Behavioral Clinical Reserach, Hollywood, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Premier Clinical Resarch Institute, Miami, Florida
  - Radiant Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Behavioral Health Hospital, Hoffman Estates, Illinois
  - Baber Research Group, Naperville, Illinois
  - Via Christi Research, Wichita, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Centerpointe Hospital, Saint Charles, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - CRI Lifetree - Marlton Unit, Marlton, New Jersey
  - Behavioral Medical Research of Brooklyn, Brooklyn, New York
  - Neurobehavioral Research, Cedarhurst, New York
  - Comprehensive Clinical Development-Queens, Jamaica, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Clinical Trials of America, Hickory, North Carolina
  - Insight Clinical Trials LLC, Shaker Heights, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Keystone Clinical Studies, Norristown, Pennsylvania
  - CRI Lifetree - Philadelphia Unit, Philadelphia, Pennsylvania
  - Berks Center for ClinicalResearch, Reading, Pennsylvania
  - Research Strategies of Memphis, Memphis, Tennessee
  - FutureSearch Clinical Trials, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Clinical Trials, L.P., Dallas, Texas
  - Pillar Clinical Research, Dallas, Texas
  - Bayou City Research, Houston, Texas
  - Alliance Research Group, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 820 subjects were screened for study participation at 53 sites in the US.
  Overall, 500 participants were included in the Safety Population: 92 rollover participants and 408 de novo participants.
Groups:
- De Novo Participants: Participants who were not part of the previous double-blind study.
  Treatment consisted of 13 subcutaneous injections of 120 mg RBP-7000 28 days apart.
  A one-time down-titration to 90 mg RBP-7000 was permitted at the investigator's discretion if the participant had tolerability issues. Participants who received the 90-mg dose of RBP-7000 and exhibited a worsening in psychiatric symptoms could receive a one-time up-titration back to 120 mg of RBP-7000 at the discretion of the investigator.
- Rollover Placebo: Participants who were randomized to the placebo arm in the double-blind study RB-US-09-0010 prior to entering this study.
  Treatment consisted of 13 subcutaneous injections of 120 mg RBP-7000 28 days apart.
  A one-time down-titration to 90 mg RBP-7000 was permitted at the investigator's discretion if the participant had tolerability issues. Participants who received the 90-mg dose of RBP-7000 and exhibited a worsening in psychiatric symptoms could receive a one-time up-titration back to 120 mg RBP-7000 at the discretion of the investigator.
- Rollover RBP-7000 90 mg: Participants who were randomized to the RBP-7000 90 mg arm in the double-blind study RB-US-09-0010 prior to entering this study.
  Treatment consisted of 11 subcutaneous injections of 120 mg RBP-7000 28 days apart (13 injections total counting the previous study).
  A one-time down-titration to 90 mg RBP-7000 was permitted at the investigator's discretion if the participant had tolerability issues. Participants who received the 90-mg dose of RBP-7000 and exhibited a worsening in psychiatric symptoms could receive a one-time up-titration back to 120 mg RBP-7000 at the discretion of the investigator.
- Rollover RBP-7000 120 mg: Participants who were randomized to the RBP-7000 120 mg arm in the double-blind study RB-US-09-0010 prior to entering this study.
  Treatment consisted of 11 subcutaneous injections of 120 mg RBP-7000 28 days apart (13 injections total counting the previous study).
  A one-time down-titration to 90 mg RBP-7000 was permitted at the investigator's discretion if the participant had tolerability issues. Participants who received the 90-mg dose of RBP-7000 and exhibited a worsening in psychiatric symptoms could receive a one-time up-titration back to 120 mg RBP-7000 at the discretion of the investigator.
Period: Overall Study
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Started | 408 | 28 | 31 | 33
Completed | 198 | 6 | 15 | 15
Not Completed | 210 | 22 | 16 | 18
Not completed — Lack of Efficacy | 7 | 0 | 1 | 1
Not completed — Adverse Event | 46 | 6 | 3 | 2
Not completed — Lost to Follow-up | 39 | 3 | 2 | 1
Not completed — Protocol Violation | 7 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 83 | 10 | 8 | 11
Not completed — Physician Decision | 27 | 0 | 2 | 3
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- De Novo Participants: Participants who were not part of the previous double-blind study.
  Treatment consisted of 13 subcutaneous injections of 120 mg RBP-7000 28 days apart.
  A one-time down-titration to 90 mg RBP-7000 was permitted at the investigator's discretion if the participant had tolerability issues. Participants who received the 90-mg dose of RBP-7000 and exhibited a worsening in psychiatric symptoms could receive a one-time up-titration back to 120 mg RBP-7000 at the discretion of the investigator.
- Total: Total of all reporting groups
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg | Total
Number analyzed (Participants) | 408 | 28 | 31 | 33 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (10.51) | 44.0 (7.33) | 41.1 (9.64) | 42.3 (10.04) | 45.1 (10.34)
Age, Customized [Count of Participants; unit: Participants]
  20 years and under | 2 | 0 | 0 | 1 | 3
  21 to 30 years | 39 | 1 | 4 | 5 | 49
  31 to 40 years | 81 | 9 | 10 | 6 | 106
  41 to 50 years | 128 | 12 | 11 | 12 | 163
  51 to 55 years | 85 | 6 | 5 | 9 | 105
  56 to 65 years | 73 | 0 | 1 | 0 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 9 | 6 | 13 | 161
  Male | 275 | 19 | 25 | 20 | 339
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 109 | 9 | 9 | 9 | 136
    Black or African American | 292 | 18 | 22 | 22 | 354
    Asian | 3 | 0 | 0 | 1 | 4
    American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 1 | 3
    Other | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 36 | 4 | 2 | 2 | 44
    Not Hispanic or Latino | 371 | 24 | 29 | 31 | 455
    Unknown | 1 | 0 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: kg] | 92.80 (20.989) | 99.33 (25.113) | 96.72 (21.305) | 94.65 (23.994) | 93.53 (21.463)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.121 (7.104) | 33.920 (8.551) | 31.926 (7.104) | 31.838 (8.341) | 31.375 (7.284)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: ratio] — A measurement of abdominal fat. Population: Measurement not taken for 10 De Novo participants.
  ratio
    number analyzed (Participants) | 398 | 28 | 31 | 33 | 490
    (all) | 0.946 (0.090) | 0.936 (0.094) | 0.975 (0.059) | 0.935 (0.075) | 0.946 (0.087)
Child-bearing Potential [Count of Participants; unit: Participants] — Population: Females only
  Participants
    number analyzed (Participants) | 133 | 9 | 6 | 13 | 161
    Yes | 54 | 4 | 3 | 5 | 66
    No | 79 | 5 | 3 | 8 | 95
Positive and Negative Syndrome Scale (PANSS) [Mean (Standard Deviation); unit: units on a scale] — The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor judgement, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 PANSS items and ranges from 30 to 210, with 30 indicating absence of symptoms of schizophrenia and 210 indicating extreme ratings of all 30 symptoms.
  units on a scale | 58.0 (8.33) | 72.9 (20.99) | 76.4 (15.99) | 71.0 (13.93) | 60.9 (12.04)
Clinical Global Impression - Severity Scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants".
  units on a scale | 3.3 (0.62) | 3.7 (1.09) | 3.8 (0.95) | 3.3 (0.89) | 3.4 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any study-related event that represents a change (positive or negative) in frequency or severity from a baseline (prestudy) event (if any), regardless of the presence of causal relationship or medical significance. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the first study dose date. AEs are determined by the Investigator to be related or not related to the study drug.
  A serious AE (SAE) is defined by federal regulation as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Although a subject may have had 2 or more adverse experiences the subject is counted only once in a category. The same subject may appear in different categories.
Time Frame: Day 1 up to week 52
Population: Safety population -- participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Number analyzed (Participants) | 408 | 28 | 31 | 33
Participants
  1 or more TEAE | 306 | 21 | 22 | 18
  >=1 TEAE related to study drug | 232 | 12 | 14 | 12
  >=1 serious TEAE | 25 | 3 | 3 | 3
  >=1 serious and related TEAE | 0 | 0 | 0 | 0
  TEAE leading to dose modification | 38 | 2 | 1 | 2
  TEAE leading to discontinuation | 47 | 6 | 3 | 2
  TEAE leading to death | 3 | 1 | 0 | 0

2. Primary Outcome: Participants With Injection Site-Related Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any study-related event that represents a change (positive or negative) in frequency or severity from a baseline (prestudy) event (if any), regardless of the presence of causal relationship or medical significance. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the first study dose date.
  Adverse events were coded using MedDRA version 17.0. Preferred terms linked to injection site AEs are reported. Although a participant may have had 2 or more AEs, the subject is counted only once in each preferred term category. The same subject may appear in different preferred term categories.
Time Frame: Day 1 up to week 52
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Number analyzed (Participants) | 408 | 28 | 31 | 33
Participants
  Injection site pain | 52 | 2 | 4 | 7
  Injection site nodule | 29 | 1 | 1 | 3
  Injection site induration | 26 | 0 | 0 | 3
  Injection site pruritus | 21 | 1 | 0 | 1
  Injection site erythema | 4 | 0 | 2 | 0
  Injection site bruising | 5 | 0 | 0 | 0
  Injection site reaction | 3 | 0 | 0 | 0
  Injection site discolouration | 1 | 0 | 0 | 1
  Injection site discomfort | 2 | 0 | 0 | 0
  Device malfunction | 2 | 0 | 0 | 0
  Implant site nodule | 1 | 0 | 0 | 0
  Influenza like illness | 1 | 0 | 0 | 0
  Infusion site bruising | 1 | 0 | 0 | 0
  Injection site irritation | 1 | 0 | 0 | 0
  Injection site swelling | 0 | 0 | 1 | 0
  Injection site ulcer | 1 | 0 | 0 | 0

3. Primary Outcome: Participants With Markedly Abnormal Weight Gain Anytime During the Study as Compared to Baseline
Description: Participants who were found to have gain >=7% and >=10% of their baseline weight at any point during the study (including unscheduled assessments) once treatment began.
Time Frame: Baseline (Day 0), Treatment (Day 1 up to Week 52)
Population: Safety population of study participants with a baseline weight recorded and at least one post-treatment weight recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Number analyzed (Participants) | 386 | 25 | 29 | 30
Participants
  >=7% increase from baseline | 106 | 3 | 4 | 5
  >=10% increase from baseline | 67 | 3 | 2 | 4

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score to Days 29, 169 and End of Study
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor judgement, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 PANSS items and ranges from 30 to 210, with 30 indicating absence of symptoms of schizophrenia and 210 indicating extreme ratings of all 30 symptoms. Negative change from baseline scores indicate improvements in symptoms.
Time Frame: Baseline (Day 0), Day 29, Day 169 and End of Study (approximately Week 52)
Population: Safety population. Population counts at each timepoint represent participants with an observation at that timepoint (all participants had baseline assessments).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Number analyzed (Participants) | 408 | 28 | 31 | 33
units on a scale
  Day 29: number analyzed (Participants) | 362 | 23 | 27 | 28
  Day 29 | -1.2 (5.70) | -4.8 (11.11) | -8.3 (13.43) | -2.4 (10.25)
  Day 169: number analyzed (Participants) | 257 | 9 | 17 | 17
  Day 169 | -1.2 (6.84) | -8.2 (18.96) | -10.0 (14.42) | -9.4 (9.62)
  End of Study: number analyzed (Participants) | 197 | 6 | 15 | 15
  End of Study | -0.4 (8.67) | -20.2 (15.59) | -12.5 (15.53) | -10.9 (13.16)

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Subscale Scores to End of Study
Description: PANSS subscales:
  * Positive scale assesses 7 items: delusions, conceptual disorganization, hallucinations, excitement, grandiosity, suspiciousness/persecution, and hostility. Scale: 7 (absent) to 49 (extreme psychopathology)
  * Negative scale assesses 7 items: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, and stereotyped thinking. Scale: 7 (absent) to 49 (extreme psychopathology)
  * General Psychopathology scale assesses 16 items: somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance. Scale: 16 (absent) to 112 (extreme psychopathology) Negative change from baseline scores indicate improvements.
Time Frame: Baseline (Day 0), End of Study (approximately Week 52)
Population: Safety population. Population counts represent participants with an end of study observation (all participants had baseline assessments).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Number analyzed (Participants) | 197 | 6 | 15 | 15
units on a scale
  Positive subscale | -1.3 (3.29) | -7.8 (5.49) | -3.7 (4.08) | -3.7 (3.50)
  Negative subscale | 1.3 (3.56) | -4.0 (5.93) | -4.1 (4.60) | -0.9 (3.78)
  General Psychopathology subscale | -0.4 (5.00) | -8.3 (6.95) | -4.7 (8.99) | -6.4 (7.92)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity Scores (CGI-S) to Days 29, 169 and End of Study
Description: The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Negative change from baseline scores indicate improvement in the severity of illness.
Time Frame: Baseline (Day 0), Baseline (Day 0), Day 29, Day 169 and End of Study (approximately Week 52)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
Number analyzed (Participants) | 408 | 28 | 31 | 33
units on a scale
  Day 29: number analyzed (Participants) | 362 | 23 | 27 | 28
  Day 29 | -0.0 (0.35) | -0.3 (0.82) | -0.2 (0.80) | -0.1 (0.71)
  Day 169: number analyzed (Participants) | 257 | 9 | 17 | 17
  Day 169 | -0.1 (0.48) | -0.3 (1.32) | -0.3 (0.59) | -0.4 (0.87)
  End of Study: number analyzed (Participants) | 197 | 6 | 15 | 15
  End of Study | -0.2 (0.66) | -1.0 (1.10) | -0.5 (0.64) | -0.3 (1.05)

ADVERSE EVENTS:
Time Frame: Day 1 to Week 52
Arm/Group | De Novo Participants | Rollover Placebo | Rollover RBP-7000 90 mg | Rollover RBP-7000 120 mg
All-Cause Mortality (participants affected / at risk) | 3/408 | 1/28 | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 25/408 | 3/28 | 3/31 | 3/33
Other Adverse Events (participants affected / at risk) | 228/408 | 14/28 | 17/31 | 13/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo Participants (N=408) | Rollover Placebo (N=28) | Rollover RBP-7000 90 mg (N=31) | Rollover RBP-7000 120 mg (N=33)
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Diverticulitus (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 4 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 5 | 1 | 0 | 1
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonany embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Substance use (Social circumstances) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | De Novo Participants (N=408) | Rollover Placebo (N=28) | Rollover RBP-7000 90 mg (N=31) | Rollover RBP-7000 120 mg (N=33)
Toothache (Gastrointestinal disorders) | 4 | 1 | 2 | 1
Fatigue (General disorders) | 12 | 1 | 3 | 1
Injection site erythema (General disorders) | 4 | 0 | 2 | 0
Injection site induration (General disorders) | 26 | 0 | 0 | 3
Injection site nodule (General disorders) | 29 | 1 | 1 | 3
Injection site pain (General disorders) | 52 | 2 | 4 | 7
Injection site pruritus (General disorders) | 21 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 8 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 23 | 1 | 2 | 0
Weight increased (Investigations) | 60 | 1 | 0 | 3
Increased appetite (Metabolism and nutrition disorders) | 16 | 0 | 1 | 2
Akathisia (Nervous system disorders) | 25 | 2 | 2 | 1
Headache (Nervous system disorders) | 20 | 0 | 4 | 1
Somnolence (Nervous system disorders) | 17 | 2 | 0 | 3
Tremor (Nervous system disorders) | 7 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 27 | 1 | 4 | 3
Schizophrenia (Psychiatric disorders) | 28 | 3 | 2 | 0
Galactorrhoea (Reproductive system and breast disorders) | 11 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multicenter publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.